CLINICAL TRIAL: NCT01415401
Title: Assessing the Efficacy and Tolerability of AZARGA® (Brinzolamide 1%/Timolol 0.5% Fixed Combination) as Replacement Therapy in Patients on COMBIGAN® (Brimonidine 0.2%/Timolol 0.5% Fixed Combination) Therapy in Canada
Brief Title: Efficacy and Tolerability of AZARGA® as Replacement Therapy in Patients on COMBIGAN® Therapy in Canada
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-11-199
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma; Ocular Hypertension; Open-angle Glaucoma
Keywords: Glaucoma; Ocular hypertension; Intraocular pressure (IOP); Open angle glaucoma; Pigment dispersion glaucoma; Pigmentary
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — brinzolamide; Timolol; Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZARGA (Experimental): Brinzolamide 1% / timolol 0.5% maleate fixed combination, 1 drop self-administered in study eye(s) twice daily for 8 weeks (8AM and 8PM)
  Interventions: Drug: Brinzolamide 1% / timolol 0.5% maleate fixed combination

INTERVENTIONS:
Drug: Brinzolamide 1% / timolol 0.5% maleate fixed combination
  Other Names: AZARGA®

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of changing to AZARGA® from prior brimonidine 0.2%/timolol 0.5% fixed combination (COMBIGAN®) therapy in patients with open-angle glaucoma or ocular hypertension and uncontrolled intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign an Informed Consent form.
* Clinical diagnosis of ocular hypertension, exfoliative open-angle or pigment dispersion glaucoma in at least one eye (study eye).
* Be on a stable IOP lowering regimen within 30 days of Screening Visit.
* IOP considered to be safe, in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Willing to discontinue the use of COMBIGAN® prior to receiving the study drug at Visit 1.
* IOP of between 19 and 35 mmHg in at least one eye (which would be the study eye) while on brimonidine/timolol fixed combination therapy.
* Best corrected visual acuity of 6/60 (20/200 Snellen, 1.0 logMAR) or better in each eye.
* Willing to follow instructions and able to attend required study visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known history of hypersensitivity to any component of the preparations used in this study.
* Presence of primary or secondary glaucoma not listed in inclusion criterion #2.
* History of ocular herpes simplex.
* Abnormality preventing reliable applanation tonometry.
* Corneal dystrophies.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye. Blepharitis or non-clinically significant conjunctival injection is allowed.
* Intraocular conventional surgery or laser surgery in study eye(s) less than 3 months prior to the Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* Women of childbearing potential not using reliable means of birth control for at least 1 month prior to the Screening/Baseline Visit.
* Pregnant or lactating.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danyel C. Carr, MS, CCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 study centers located in Canada.
Pre-assignment Details: Of the 57 enrolled, 3 participants were exited as screen failures. This reporting group includes all participants who received study medication (54).
Period: Overall Study
Arm/Group | AZARGA
Started | 54
Completed | 47
Not Completed | 7
Not completed — Adverse Event | 5
Not completed — DId not meet inclusion/exclusion criteri | 1
Not completed — Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who received study medication.
Arm/Group | AZARGA
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in IOP at the Final Visit From Prior Brimonidine 0.2%/Timolol 0.5% Fixed Combination (COMBIGAN®) Therapy (i.e. From Baseline)
Description: IOP (fluid pressure inside the eye) was assessed by Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Baseline, Week 8
Population: This analysis population includes all subjects who received study medication and had at least one on-therapy study visit. Last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZARGA
Number analyzed (Participants) | 54
mmHg
  Baseline | 22.24 (3.150)
  Change from baseline at Week 8 | -2.24 (3.928)

2. Secondary Outcome: Percentage of Subjects Who Reach Target IOP (≤ 18 mmHg)
Description: IOP (fluid pressure inside the eye) was assessed by Goldmann applanation tonometry and measured in mmHg. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Week 8
Population: This analysis population includes all subjects who received study medication, completed all study visits, and satisfied inclusion/exclusion criteria. In addition, no imputation methods were employed; therefore only efficacy measurements available at each visit and time point were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | AZARGA
Number analyzed (Participants) | 47
percentage of participants | 36.2

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (1 year, 9 months). This analysis group includes all subjects who received study medication.
Description: An AE is defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Adverse events were obtained as solicited comments from the study patients and as observations by the Investigator as outlined in the study protocol.
Arm/Group | AZARGA
Serious Adverse Events (participants affected / at risk) | 1/54
Other Adverse Events (participants affected / at risk) | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZARGA (N=54)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.